CLINICAL TRIAL: NCT02816346
Title: Dose-Finding Study of Lyophilized Shigella Sonnei 53G Challenge Strain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VAC-048
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: shigella
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: target dose of 500 CFU (Experimental): Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Received target dose of 500 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 510, 717, 588, and 567 CFU).
  Interventions: Biological: Shigella sonnei 53G
- Cohort 2: target dose of 1000 CFU (Experimental): Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Received target dose of 1000 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 817 CFU), since the attack rate of shigellosis for Cohort 1 was below the protocol target of 60%.
  Interventions: Biological: Shigella sonnei 53G
- Cohort 3: target dose of 1000 CFU (Experimental): Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Received target dose of 1000 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 913 CFU. Although the target dose was the same as Cohort 2, the safety monitoring committee felt that the per-protocol a priori definition of shigellosis was too restrictive and that increasing the dose above 1000 CFU may lead to unnecessarily high toxicity.
  Interventions: Biological: Shigella sonnei 53G
- Cohort 4: target dose of 1500 CFU (Experimental): Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Received target dose of 1500 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 1760 CFU) since the attack rate of shigellosis for Cohort 2 and 3 was below the protocol target of 60%.
  Interventions: Biological: Shigella sonnei 53G
- Cohort 5: target dose of CFU (Experimental): Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Received target dose of 1150 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 1760 CFU) as the final confirmatory cohort since it was felt that the disease rate and profile of Cohort 4 was appropriate.
  Interventions: Biological: Shigella sonnei 53G

INTERVENTIONS:
Biological: Shigella sonnei 53G — Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)

SUMMARY:
Development of an S. sonnei human challenge model using a newly manufactured lyophilized lot of S. sonnei strain 53G (Lot 1794) that can be used in the future as a challenge strain for all S. sonnei vaccine candidates. An adaptable dosing plan was used to determine the dose of Shigella sonnei 53G that induces the primary outcome in approximately 60% of subjects.

DETAILED DESCRIPTION:
Primary objectives:

1. Establish a human challenge model of S. sonnei 53G infection using a lyophilized formulation of the challenge strain.
2. Identify a dose of lyophilized S. sonnei 53G that induces the primary outcome in approximately 60% of subjects with no adverse safety concerns.

Secondary objectives:

1. Estimate quantitative shedding and basic immunogenicity of the challenge strain.
2. Collect and archive blood and fecal samples for systems biology, microbiome, and other omics-based work to be conducted under a separate research protocol in future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female between 18 and 49 years of age (inclusive).
2. General good health defined as (a) no significant medical illness, (b) no clinically significant physical examination findings and (c) no screening laboratory values significantly outside the normal limits of the testing laboratory within 45 days of challenge.
3. Demonstrate comprehension of the protocol procedures and knowledge of study by passing a written examination (pass grade ≥70%) on day -1.
4. Willing to sign an informed consent form (ICF).
5. Willingness to participate for an inpatient stay lasting up to 11 days and an outpatient follow-up lasting 6 months from challenge.
6. Willing to not smoke during the inpatient stay.
7. Available for all planned follow-up visits.
8. Negative serum pregnancy test at screening and negative urine pregnancy test on the day of admission to the inpatient phase for female subjects of childbearing potential. Females of childbearing potential must agree to use an effective method of birth control (birth control pills, injection hormonal contraceptive, implant hormonal contraceptive,

   hormonal patch, intrauterine device (IUD), sterilization by hysterectomy or tubal ligation, spermicidal products and barrier methods such as cervical sponge, diaphragm, or condom) within two months of challenge and during the entire study. Abstinence is acceptable. A woman is eligible if she is monogamous with a vasectomized partner.
9. Willing to not donate blood for up to 6 months after completion of the inpatient phase of the study.
10. Willing to refrain from participation in another investigational vaccine or drug trial at least until after completion of the 6 month follow-up safety call.

Exclusion Criteria:

1. Presence of a significant medical condition (e.g. psychiatric conditions, alcohol or illicit drug abuse/dependency, or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
2. Immunosuppressive illness or immunoglobulin A (IgA) deficiency
3. Positive serology results for HIV, HBsAg, hepatitis C virus (HCV), or syphilis (RPR) antibodies.
4. Evidence of inflammatory arthritis on exam and/or human leukocyte antigen B27 (HLA-B27) positive.
5. Family history of inflammatory arthritis.
6. Significant abnormalities in screening lab hematology or serum chemistry, as determined by PI.
7. Allergy to fluoroquinolones or trimethoprim-sulfamethoxazole
8. Fewer than 3 stools per week or more than 3 stools per day as the usual frequency.
9. History of diarrhea in the 2 weeks prior to planned inpatient phase
10. Use of antibiotics during the 7 days before receiving the challenge inoculum dosing
11. Use of prescription and/or over the counter (OTC) medications that contain Imodium, acetaminophen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs, during the 48 hours prior to investigational product administration
12. Travel within two years prior to dosing to countries where Shigella infection is endemic.
13. Use of any medication known to affect the immune function [e.g., oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent and others): nasal and topical steroids are allowed] within 30 days preceding receipt of the challenge inoculum or planned use during the active study period.
14. Serologic evidence of Shigella sonnei (titer > 1:2500)
15. A positive urine test for opiates.
16. A chronic disease (such as hypertension, hyperlipidemia or anxiety/depression) for which doses of prescription medications are not stable for at least the past 3 months.
17. Scheduled and/or long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal, intra-articular, and topical steroids are allowed)
18. Have immunocompromised household contacts.
19. A clinically significant abnormality on physical examination, including a systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg, or a resting pulse >100 beats/min or <55 beats/min (<50 beats/min for conditioned athletes).
20. Pregnant, nursing, or plan to become pregnant within 6 months of receipt of the study product.
21. In the 4 weeks following challenge, subject will be living with or having daily contact with elderly persons aged 70 years or more, diapered individuals, persons with disabilities, children <2 years old, or a woman known to be pregnant or nursing, or anyone with diminished immunity. This includes contact at home, school, day-care, nursing homes, or similar places.
22. Work in a health care setting, day care center, or as a food handler in the 4 weeks following the challenge with S. sonnei.
23. Use of any investigational drug or any investigational vaccine within 60 days preceding challenge, or planned use during the 6 months after receipt of the study agent.
24. Have received a licensed, live vaccine within 28 days or a licensed inactivated vaccine within 14 days of receiving the challenge inoculum.
25. Inability to comply with inpatient rules and regulations.
26. Has any other condition that, in the opinion of the Investigator, would jeopardize the safety or rights of a participant or would render the subject unable to comply with the protocol.
27. Received blood or blood products within the past six months.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-09-12; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frenck, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liechty Z, Baldwin A, Isidean S, Suvarnapunya A, Frenck R, Porter C, Goodson M. Dynamics of the gut microbiome in subjects challenged with Shigella sonnei 53G in a controlled human infection model. mSphere. 2025 Apr 29;10(4):e0090624. doi: 10.1128/msphere.00906-24. Epub 2025 Mar 28. PMID 40152601

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the recruiting range of Cincinnati Children's Hospital Medical Center (CCHMC) via word of mouth and advertisements in multiple formats including but not limited to newspapers, fliers, e-mails, and the CCHMC website.
Groups:
- Cohort 1: S. Sonnei 53G Target Dose 500 CFU: Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Target Dose: 500cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 2: S. Sonnei 53G Target Dose 1000 CFU: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 1 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Dose: 1000 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 3: S. Sonnei 53G Target Dose of 1000 CFU: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 2 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Dose: 1000 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 4: S. Sonnei 53G Target Dose 1500 CFU: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 3 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Dose: 1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 5: S. Sonnei 53G Target Dose 1150 CFU: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 4 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: One dose of Shigella sonnei rehydrated challenge strain 53G (Lot 1794) suspension in 2 mL of cold sterile water combined and diluted in cold, sterile normal saline 0.9% (i.e. challenge suspension).
  Mode of Administration: After a 90 minute fast subjects will drink the 120 mL of sodium bicarbonate (to neutralize gastric acidity) and then drink the challenge suspension within 5 minutes.
  Dose: 1150 cfu (doses were to be increased or lowered based on results of preceding cohorts)
Period: Overall Study
Arm/Group | Cohort 1: S. Sonnei 53G Target Dose 500 CFU | Cohort 2: S. Sonnei 53G Target Dose 1000 CFU | Cohort 3: S. Sonnei 53G Target Dose of 1000 CFU | Cohort 4: S. Sonnei 53G Target Dose 1500 CFU | Cohort 5: S. Sonnei 53G Target Dose 1150 CFU
Started | 10 | 10 | 10 | 10 | 16
Completed | 10 | 10 | 10 | 10 | 16
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Received 500 colony-forming units (CFU) of Shigella sonnei 53G.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 2: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 1 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 3: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 2 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 4: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 3 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 5: Received higher dose of Shigella sonnei 53G if ≥ 60% of subjects in Cohort 4 experienced shigellosis, or lower dose if not.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16 | 56
Age, Continuous [Geometric Mean (Standard Deviation); unit: years] | 35.7 (10.7) | 32.3 (9.9) | 34.3 (9.9) | 32.2 (8.8) | 30.1 (8.8) | 32.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 6 | 7 | 10 | 33
  Male | 3 | 7 | 4 | 3 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 10 | 10 | 16 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 10 | 10 | 14 | 52
  White | 1 | 0 | 0 | 0 | 2 | 3
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Shigellosis
Description: Per protocol definition: shedding of S. sonnei in the stool accompanied by moderate-severe diarrhea (4 or more loose/watery Grade 3-5 stools or 400+ gram stools per 24 hours, or requires medical intervention) and/or dysentery (a Grade 3, 4, or 5 stool with gross blood on at least 2 occasions and reportable constitutional symptoms) along with moderate fever (Oral temperature of ≥101.2°F) or one or more severe intestinal symptoms.
  Alternative endpoint 1 definition: severe diarrhea, or moderate diarrhea plus fever, or moderate diarrhea plus 1 moderate constitutional/enteric symptom, or dysentery.
  Alternative endpoint 2 definition: severe diarrhea, or moderate diarrhea plus fever, or moderate diarrhea plus 1 severe constitutional/enteric symptom, or dysentery plus 1 severe constitutional/enteric symptom
Time Frame: 11 days after administration of S. sonnei
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Received target dose of 500 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 510, 717, 588, and 567 CFU).
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 2: Received target dose of 1000 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 817 CFU), since the attack rate of shigellosis for Cohort 1 was below the protocol target of 60%.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 3: Received target dose of 1000 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 913 CFU. Although the target dose was the same as Cohort 2, the safety monitoring committee felt that the per-protocol a priori definition of shigellosis was too restrictive and that increasing the dose above 1000 CFU may lead to unnecessarily high toxicity.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 4: Received target dose of 1500 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 1760 CFU) since the attack rate of shigellosis for Cohort 2 and 3 was below the protocol target of 60%.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
- Cohort 5: Received target dose of 1150 colony-forming units (CFU) of Shigella sonnei 53G (actual dose: 1760 CFU) as the final confirmatory cohort since it was felt that the disease rate and profile of Cohort 4 was appropriate.
  Shigella sonnei 53G: Investigational Product: Shigella sonnei strain 53G (Lot 1794) Mode of Administration: Delivered with sodium bicarbonate orally after a 90 minute fast.
  Dose: 500-1500 cfu (doses were to be increased or lowered based on results of preceding cohorts)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
Participants
  Per protocol definition: Yes | 0 | 2 | 1 | 4 | 2
  Per protocol definition: No | 10 | 8 | 9 | 6 | 14
  Alternative endpoint 1: Yes | 0 | 6 | 4 | 7 | 7
  Alternative endpoint 1: No | 10 | 4 | 6 | 3 | 9
  Alternative endpoint 2: Yes | 0 | 5 | 3 | 6 | 7
  Alternative endpoint 2: No | 10 | 5 | 7 | 4 | 9

2. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Stool: Lipopolysaccharide (LPS) Antigen
Description: IgA (total and S. sonnei specific) will be determined in fecal extracts using standard ELISA. IgA was recovered from stool samples using a soybean trypsin inhibitor ethylenediaminetetraacetic acid (EDTA) procedure. The shigella-antigen specific activity was calculated by dividing the endpoint titer by the IgA concentration in matched samples.
Time Frame: Baseline (days -5,-1), Day 3, Day 7, and Day 14
Population: Stool samples were not collected from all subjects at all time points. Samples containing less than 2 ug/mL of total IgA were excluded from analysis. If both baseline samples were below 2 ug/mL, the subject was excluded from analysis.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline 1 (Day -5): number analyzed (Participants) | 10 | 6 | 9 | 4 | 11
  Baseline 1 (Day -5) | 19 (130) | 11 (8) | 11 (24) | 17 (157) | 8 (6)
  Baseline 2 (Day -1): number analyzed (Participants) | 10 | 8 | 9 | 10 | 10
  Baseline 2 (Day -1) | 15 (53) | 8 (26) | 11 (51) | 9 (200) | 10 (15)
  Day 3 | 15 (65) | 11 (14) | 9 (11) | 11 (99) | 11 (21)
  Day 7: number analyzed (Participants) | 10 | 10 | 9 | 10 | 16
  Day 7 | 49 (121) | 70 (413) | 80 (136) | 49 (296) | 42 (155)
  Day 14: number analyzed (Participants) | 10 | 9 | 10 | 9 | 16
  Day 14 | 211 (1024) | 40 (841) | 226 (371) | 101 (205) | 57 (431)

3. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Stool: Invaplex Antigen
Description: IgA (total and S. sonnei specific) will be determined in fecal extracts using standard ELISA. IgA was recovered from stool samples using a soybean trypsin inhibitor-EDTA procedure. The shigella-antigen specific activity was calculated by dividing the endpoint titer by the IgA concentration in matched samples.
Time Frame: Baseline (days -5,-1), Day 3, Day 7, and Day 14
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline 1 (Day -5): number analyzed (Participants) | 10 | 6 | 9 | 3 | 11
  Baseline 1 (Day -5) | 20 (211) | 18 (60) | 10 (104) | 20 (638) | 11 (22)
  Baseline 2 (Day -1): number analyzed (Participants) | 10 | 8 | 9 | 10 | 10
  Baseline 2 (Day -1) | 19 (130) | 12 (111) | 9 (105) | 10 (403) | 9 (11)
  Day 3 | 19 (130) | 15 (98) | 6 (2) | 16 (400) | 80 (441)
  Day 7: number analyzed (Participants) | 10 | 10 | 9 | 10 | 16
  Day 7 | 53 (140) | 92 (381) | 50 (124) | 80 (441) | 84 (498)
  Day 14: number analyzed (Participants) | 10 | 10 | 10 | 9 | 16
  Day 14 | 422 (3317) | 118 (1679) | 320 (459) | 403 (540) | 104 (478)

4. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Description: Blood (10 mL) was collected on days -1, 7, 14, 28 and 56 for Immunoglobulin A (IgA), Immunoglobulin M (IgM), and Immunoglobulin G (IgG) assay by Enzyme linked immunosorbent assay (ELISA).
Time Frame: 57 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline (Day -1) | 528 (611) | 492 (547) | 246 (450) | 459 (420) | 497 (3137)
  Day 7 | 746 (913) | 919 (3813) | 400 (458) | 857 (1315) | 951 (6276)
  Day 14 | 4222 (19953) | 2425 (7591) | 6859 (15472) | 3676 (9816) | 3200 (17160)
  Day 28 | 2425 (15506) | 1715 (8165) | 3430 (15370) | 1715 (4974) | 1532 (6991)
  Day 56 | 1393 (3897) | 1131 (8350) | 1372 (2418) | 1300 (4188) | 1131 (12550)

5. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Serum: Lipopolysaccharide (LPS) Antigen
Description: as for outcome 4
Time Frame: 57 days
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline (Day -1) | 373 (666) | 264 (610) | 123 (138) | 348 (2073) | 248 (823)
  Day 7 | 528 (611) | 1213 (10390) | 264 (344) | 919 (2474) | 1037 (3047)
  Day 14 | 4222 (16541) | 2425 (10086) | 3200 (9864) | 2111 (7898) | 3644 (10457)
  Day 28 | 2425 (15598) | 857 (5990) | 919 (2444) | 919 (4032) | 1288 (4164)
  Day 56 | 919 (877) | 528 (1212) | 635 (1219) | 800 (2532) | 591 (1784)

6. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin G (IgG) Antibodies in Serum: Invaplex Antigen
Description: as for outcome 4
Time Frame: 57 days
Population: No sample was available for one subject in Cohort 3 on Day 56.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline (Day -1) | 2599 (5412) | 2599 (1960) | 2986 (15270) | 2263 (4011) | 1745 (12365)
  Day 7 | 3430 (7619) | 3940 (4221) | 3200 (7303) | 3940 (3477) | 3490 (24798)
  Day 14 | 10397 (31301) | 7352 (30508) | 14703 (14347) | 11143 (18203) | 8300 (28740)
  Day 28 | 9701 (18863) | 6859 (14595) | 11943 (14904) | 9701 (9361) | 6683 (33105)
  Day 56: number analyzed (Participants) | 10 | 10 | 9 | 10 | 16
  Day 56 | 6400 (9199) | 4525 (7013) | 10159 (9659) | 5971 (4758) | 4525 (16370)

7. Secondary Outcome: Geometric Mean Titer (GMT) of Immunoglobulin A (IgA) Antibodies in Serum: Invaplex Antigen
Description: as for outcome 4
Time Frame: 57 days
Population: No sample was available for one subject in Cohort 3 on Day 56.
Measure: Geometric Mean (Standard Deviation); unit: titer
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 16
titer
  Baseline (Day -1) | 348 (596) | 283 (330) | 115 (113) | 400 (3957) | 183 (1694)
  Day 7 | 429 (451) | 1056 (4076) | 528 (420) | 1600 (8146) | 1131 (3217)
  Day 14 | 3200 (16194) | 2263 (7995) | 5198 (7205) | 7879 (19368) | 5620 (13385)
  Day 28 | 1970 (4825) | 1213 (4011) | 1715 (3660) | 2425 (7953) | 1822 (4613)
  Day 56 | 985 (1046) | 650 (1180) | 864 (2032) | 1213 (5145) | 872 (2105)

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/16
Other Adverse Events (participants affected / at risk) | 6/10 | 10/10 | 10/10 | 10/10 | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=10) | Cohort 2 (N=10) | Cohort 3 (N=10) | Cohort 4 (N=10) | Cohort 5 (N=16)
Abdominal Pain (Gastrointestinal disorders) | 1 | 9 | 7 | 7 | 9
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 11
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2 | 2 | 1
Asthma (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Bacterial vaginosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 3 | 2 | 1 | 3
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure systolic decreased (Investigations) | 0 | 0 | 0 | 0 | 6
Blood pressure systolic increased (Investigations) | 0 | 4 | 10 | 5 | 6
Blood sodium increased (Investigations) | 0 | 0 | 2 | 0 | 0
Bowel movement irregularity (Investigations) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Chills (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 7 | 7 | 12
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Ear infection (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 3 | 2 | 4 | 4
Haemorrhoids (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 7 | 8 | 7 | 10
Heart rate decreased (Investigations) | 0 | 1 | 0 | 0 | 2
Heart rate increased (Investigations) | 0 | 2 | 4 | 7 | 6
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 1 | 1 | 2
Neutrophil count increased (Investigations) | 0 | 2 | 0 | 3 | 0
Oropharyngeal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Swelling face (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 1 | 1 | 3
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 1 | 1 | 3
White blood cell count increased (Investigations) | 0 | 2 | 2 | 2 | 0
Not recorded (General disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 3 | 3 | 4
Gas (Gastrointestinal disorders) | 1 | 8 | 5 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 7 | 7 | 3 | 5
Malaise (General disorders) | 0 | 8 | 8 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 9 | 2 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 7 | 1 | 3 | 1
Fever (General disorders) | 0 | 3 | 1 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT02816346/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT02816346/SAP_001.pdf